CLINICAL TRIAL: NCT01847222
Title: An Assessment of the Safety and Pharmacokinetics of Ascending Doses of SANGUINATE™ in Healthy Volunteers.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to completion of competing study.
Sponsor: Prolong Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SGHV-005
Record Dates: First submitted 2013-04-23; First posted 2013-05-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Drug Safety
MeSH Terms: interventions — PEGylated carboxyhemoglobin bovine; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- SANGUINATE™ (Experimental): PEG-bHb-CO
  Interventions: Biological: SANGUINATE™
- Normal Saline Solution (Placebo Comparator): Saline Solution
  Interventions: Drug: Normal Saline Solution

INTERVENTIONS:
Biological: SANGUINATE™ — PEG-bHb-CO
  Other Names: PEG-bHb-CO
  Arms: SANGUINATE™
Drug: Normal Saline Solution — Placebo
  Other Names: Placebo
  Arms: Normal Saline Solution

SUMMARY:
Safety assessment of SANGUINATE™ in Healthy Volunteers.

DETAILED DESCRIPTION:
Safety and Pharmacokinetic assessment in ascending doses of SANGUINATE™ in Healthy Volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male Volunteers;
* Age ≥18 years and ≤45 years;
* BMI ≥20- ≤30 kg/m²
* No clinically significant screening observations

Exclusion Criteria:

* Female volunteers;
* Any history of significant cardiac, renal, neurologic, metabolic, pulmonary, gastrointestinal, chronic hepatic disease or any other disease which in the judgment of the Investigator would interfere with the study or confound the results;
* History of allergy or major allergic reactions considered to be clinically significant by the Investigator;
* Any screening assessment determined to be clinically significant by the Investigator;
* Donate blood within 60 days of screening or otherwise experienced blood loss >250 mL within the same period;

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability. | 7 days
  Adverse events of SANGUINATE™

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Brenner, MD, Principal Investigator — Rambam Health Care Facility
Locations (1):
- Rambam Health Care Facility, Haifa, Israel